CLINICAL TRIAL: NCT01490086
Title: REFRESH : Randomized Double-blind, Placebo-controlled, Multicenter Trial to Assess the Safety and Efficacy of RP5063 in Subjects With an Acute Exacerbation of Schizophrenia or Schizoaffective Disorder
Brief Title: RP5063 in Subjects With Schizophrenia or Schizoaffective Disorder
Acronym: REFRESH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Reviva Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RVP-20-001
Record Dates: First submitted 2011-12-07; First posted 2011-12-12 (Estimated); Results first posted 2015-01-26 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Acute Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Psychotic Disorders | interventions — RP5063; Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 15 mg RP5063 daily (Experimental): RP5063 15 mg once daily
  Interventions: Drug: RP5063
- 30 mg RP5063 daily (Experimental): RP5063 30 mg once daily
  Interventions: Drug: RP5063
- 50 mg RP5063 daily (Experimental): RP5063 50 mg once daily
  Interventions: Drug: RP5063
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: placebo
- aripiprazole (Active Comparator): aripiprazole 15 mg daily
  Interventions: Drug: aripiprazole

INTERVENTIONS:
Drug: RP5063 — daily
  Arms: 15 mg RP5063 daily; 30 mg RP5063 daily; 50 mg RP5063 daily
Drug: placebo — daily
  Arms: Placebo
Drug: aripiprazole — daily
  Other Names: Abilify
  Arms: aripiprazole

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of RP5063 relative to placebo for the treatment of schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients providing informed consent prior to any study specific procedures
* Patients meeting Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for schizophrenia (paranoid type, disorganized type, catatonic type or undifferentiated type), or schizoaffective disorder
* Patients with normal physical examination, laboratory, vital signs,and electrocardiogram (ECG)

Exclusion Criteria:

* Patients with other primary psychiatric disorders as delirium, or bipolar I or II disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2011-12; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M Cantillon, Study Director — Fundacion REVIVA, Red de VIH del Valle del Cauca
Locations (15):
- Reviva site, Philadelphia, Pennsylvania, United States
- India (7):
  - Reviva site, Bangalore
  - Reviva site, Chennai
  - Reviva site, Guntur
  - Reviva site, Jaipur
  - Reviva site, Kanpur
  - Reviva site, Lucknow
  - Reviva site, Mangalore
- Malaysia (3):
  - Reviva site, Johor Bahru
  - Reviva site, Kuala Lumpur
  - Reviva Site, Tanjung Rambutan
- Reviva site, Chisinau, Moldova
- Philippines (3):
  - Reviva site, Mandaluyong
  - Reviva site, Mandurriao
  - Reviva site, Subandaku

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 270 Subjects with acute exacerbation Schizophrenia and Schizoaffective disorder were selected from multiple sites in USA, Moldova, India, Philippines and Malaysia between December 2011 and January 2013.
Pre-assignment Details: Subjects were screened over a period of 7 days in the site's in-patient facility. 270 subjects were recruited. Of these, 36 subjects did not meet the study eligibility criteria. Therefore, a total of 234 subjects were enrolled into the study.
Groups:
- RP5063 15 mg: Participants with acute schizophrenia or schizoaffective disorder receiving 15 mg of RP5063 once daily for 28 days.
- RP5063 30 mg: Participants with acute schizophrenia or schizoaffective disorder receiving 30 mg of RP5063 once daily for 28 days.
- RP5063 50 mg: Participants with acute schizophrenia or schizoaffective disorder receiving 50 mg of RP5063 once daily for 28 days.
- Aripiprazole 15 mg: Participants with acute schizophrenia or schizoaffective disorder receiving 15 mg of Aripiprazole once daily for 28 days.
- Placebo: Participants with acute schizophrenia or schizoaffective disorder receiving Placebo once daily for 28 days.
Period: Overall Study
Arm/Group | RP5063 15 mg | RP5063 30 mg | RP5063 50 mg | Aripiprazole 15 mg | Placebo
Started | 58 | 59 | 58 | 20 | 39
Completed | 50 | 44 | 51 | 13 | 28
Not Completed | 8 | 15 | 7 | 7 | 11
Not completed — Consent withdrawn | 4 | 4 | 3 | 0 | 1
Not completed — Non-compliance | 0 | 1 | 0 | 0 | 0
Not completed — Abnormal laboratory findings | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 3 | 4 | 2 | 3 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0
Not completed — Lack of Efficacy | 0 | 3 | 1 | 0 | 8
Not completed — Worsening of symptoms | 0 | 1 | 0 | 1 | 0
Not completed — Subject uncontrollable and abusive | 0 | 1 | 0 | 0 | 0
Not completed — Subject left hospital | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population is the Safety Population (Total 233), which comprises all enrolled subjects (Total 234) who received at least one dose of study treatment. One Placebo subject was enrolled in the study but did not receive any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | RP5063 15 mg | RP5063 30 mg | RP5063 50 mg | Aripiprazole 15 mg | Placebo | Total
Number analyzed (Participants) | 58 | 59 | 58 | 20 | 38 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (10) | 37 (12) | 35 (9) | 35 (10) | 36 (12) | 36 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 16 | 2 | 11 | 55
  Male | 41 | 50 | 42 | 18 | 27 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 58 | 59 | 58 | 20 | 37 | 232
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 51 | 53 | 52 | 18 | 34 | 208
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 1 | 1
  Black or African American | 3 | 3 | 3 | 1 | 1 | 11
  White | 3 | 3 | 3 | 1 | 2 | 12
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 1 | 2 | 12
  Philippines | 15 | 15 | 15 | 5 | 9 | 59
  Malaysia | 10 | 11 | 10 | 3 | 8 | 42
  Moldova, Republic of | 3 | 3 | 3 | 1 | 2 | 12
  India | 27 | 27 | 27 | 10 | 17 | 108

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Schizophrenia Symptoms: Positive and Negative Syndrome Scale (PANSS) Total Score
Description: PANSS total score comprises Positive (Delusions, Conceptual disorganization, Hallucinatory behavior, Excitement, Grandiosity, Suspiciousness/persecution, Hostility), Negative (Blunted affect, Emotional withdrawal, Poor rapport, Passive/apathetic social withdrawal, Difficulty in abstract thinking, Lack of spontaneity and flow of conversation, Stereotyped thinking), and General Psychopathology (Somatic concern, Anxiety, Guilt feelings, Tension, Mannerisms and posturing, Depression, Motor retardation, Uncooperativeness, Unusual thought content, Disorientation, Poor attention, Lack of judgment and insight, Disturbance of volition, Poor impulse control, Preoccupation, Active social avoidance) Scales. Scores are obtained by adding the ratings of each item in each scale. Range is 7-49 for Positive and Negative scores; 16-112 for General Psychopathology score; and 30-210 for Total score. Higher score reflects worse outcome; larger reduction from baseline reflects better outcome.
Time Frame: Baseline to Day 28
Population: The ITT population is comprised of participants who had received at least one dose of treatment, have baseline and at least one assessment of PANSS and CGI-S without major deviations at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | RP5063 15 mg | RP5063 30 mg | RP5063 50 mg | Aripiprazole 15 mg | Placebo
Number analyzed (Participants) | 56 | 57 | 57 | 19 | 37
scores on a scale
  Baseline | 87.57 (13.30) | 88.74 (13.37) | 85.88 (14.86) | 91.68 (16.10) | 89.84 (15.60)
  Day 28 | 67.34 (21.98) | 73.32 (20.24) | 66.67 (19.66) | 82.37 (22.13) | 78.43 (24.14)

2. Secondary Outcome: Demonstrates Antipsychotic Efficacy as Assessed by Change From Baseline on the Clinical Global Impression Scale - Severity (CGI-S)
Description: Clinical Global Impression, Severity (CGI-S) is a single-item (7-point) scale that evaluates the overall severity of the subject's mental illness. Scores range from 1 (not ill at all) to 7 (among the most extremely ill). A reduction in score indicates an improvement in the subject's condition.
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | RP5063 15 mg | RP5063 30 mg | RP5063 50 mg | Aripiprazole 15 mg | Placebo
Number analyzed (Participants) | 56 | 57 | 57 | 19 | 37
scores on a scale
  Baseline | 4.79 (0.56) | 4.81 (0.77) | 4.75 (0.71) | 4.84 (0.60) | 4.76 (0.55)
  Day 28 | 3.48 (1.22) | 3.93 (1.24) | 3.54 (1.05) | 4.53 (1.02) | 4.05 (1.27)

3. Secondary Outcome: Demonstrates Antipsychotic Efficacy as Assessed by Change From Baseline on the PANSS Positive Subscale
Description: The Positive Scale includes 7 Items (Delusions, Conceptual disorganization, Hallucinations, Hyperactivity, Grandiosity, Suspiciousness/persecution, Hostility) and is calculated by adding the subscale item scores to obtain results ranging from 7 to 49. A higher score reflects worse outcome and a larger reduction in the score from baseline reflects better treatment efficacy.
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | RP5063 15 mg | RP5063 30 mg | RP5063 50 mg | Aripiprazole 15 mg | Placebo
Number analyzed (Participants) | 56 | 57 | 57 | 19 | 37
scores on a scale
  Baseline | 24.79 (4.21) | 23.77 (4.66) | 23.68 (4.73) | 25.42 (6.77) | 24.54 (3.78)
  Day 28 | 17.82 (7.95) | 18.75 (7.27) | 16.72 (6.66) | 23.47 (7.88) | 19.95 (6.84)

4. Secondary Outcome: Demonstrates Antipsychotic Efficacy as Assessed by Change From Baseline on the PANSS Negative Subscale
Description: The Negative Scale includes 7 items (Blunted affect, Emotional withdrawal, Poor rapport, Passive/apathetic social withdrawal, Difficulty in abstract thinking, Lack of spontaneity and flow of conversation, Stereotyped thinking) and is calculated by adding the negative subscale item scores to obtain results ranging from 7 to 49. Minimum score is 7, maximum score is 49. A higher score reflects worse outcome and a larger reduction in the score from baseline reflects better treatment efficacy.
Time Frame: Baseline to Day 28
Population: The ITT population is comprised of participants who had receiving at least one dose of treatment, have baseline and at least one assessment of PANSS and CGI-S without major deviations at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | RP5063 15 mg | RP5063 30 mg | RP5063 50 mg | Aripiprazole 15 mg | Placebo
Number analyzed (Participants) | 56 | 57 | 57 | 19 | 37
scores on a scale
  Baseline | 21.80 (5.63) | 22.89 (5.25) | 21.37 (5.91) | 22.53 (4.38) | 22.24 (6.34)
  Day 28 | 16.96 (5.11) | 19.21 (5.92) | 17.72 (5.89) | 19.47 (5.16) | 20.57 (6.64)

5. Secondary Outcome: Demonstrates Antipsychotic Efficacy as Assessed by Change From Baseline on the PANSS General Psychopathology Subscale
Description: The General Psychopathology Scale consists of 16 items (Somatic concern, Anxiety, Guilt feelings, Tension, Mannerisms and posturing, Depression, Motor retardation, Uncooperativeness, Unusual thought content, Disorientation, Poor attention, Lack of judgment and insight, Disturbance of volition, Poor impulse control, Preoccupation, Active social avoidance). The General Psychopathology score is obtained by adding the ratings of each item in the scale, with results ranging from 16 to 112. A higher score reflects worse outcome and a larger reduction in the score from baseline reflects better treatment efficacy.
Time Frame: Baseline to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | RP5063 15 mg | RP5063 30 mg | RP5063 50 mg | Aripiprazole 15 mg | Placebo
Number analyzed (Participants) | 56 | 57 | 57 | 19 | 37
scores on a scale
  Baseline | 40.98 (7.30) | 42.07 (7.08) | 40.82 (7.61) | 43.74 (9.41) | 43.05 (8.36)
  Day 28 | 32.55 (11.26) | 35.35 (10.12) | 32.23 (9.79) | 39.42 (11.25) | 37.92 (13.03)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over a period of 14 months.
Description: All subjects receiving at least one dose of investigational product were included in the safety analyses. A total of 233 subjects out of randomized 234 subjects were exposed to the investigational product, provided post-baseline safety data and were included in the safety population.
Arm/Group | RP5063 15 mg | RP5063 30 mg | RP5063 50 mg | Aripiprazole 15 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/58 | 1/59 | 1/58 | 2/20 | 0/38
Other Adverse Events (participants affected / at risk) | 29/58 | 30/59 | 37/58 | 10/20 | 23/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RP5063 15 mg (N=58) | RP5063 30 mg (N=59) | RP5063 50 mg (N=58) | Aripiprazole 15 mg (N=20) | Placebo (N=38)
Elevated liver enzyme levels (Investigations) | 1 | 1 | 1 | 1 | 0
Sedation excessive (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RP5063 15 mg (N=58) | RP5063 30 mg (N=59) | RP5063 50 mg (N=58) | Aripiprazole 15 mg (N=20) | Placebo (N=38)
Tachycardia (Cardiac disorders) | 0 | 1 | 2 | 1 | 0
Hyperprolactinaemia (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Oculogyric crisis (Eye disorders) | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 3 | 1 | 2
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 2 | 1 | 1 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Akathisia (Nervous system disorders) | 1 | 3 | 6 | 0 | 0
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 2 | 3 | 5 | 1 | 0
Headache (Nervous system disorders) | 3 | 1 | 2 | 1 | 1
Sedation (Nervous system disorders) | 0 | 0 | 2 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 3 | 0 | 0
Tremor (Nervous system disorders) | 1 | 3 | 2 | 0 | 1
Affective disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0
Agitation (Psychiatric disorders) | 6 | 6 | 4 | 4 | 6
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 16 | 15 | 10 | 4 | 8
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Restlessness (Psychiatric disorders) | 1 | 3 | 2 | 1 | 3
Schizophrenia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Social avoidant behavior (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less